CLINICAL TRIAL: NCT06341998
Title: Clinical Study of Sirolimus Combined With Chemotherapy in the Treatment of Recurrent/Refractory Yolk Sac Tumor in Children
Brief Title: Clinical Study of Chemotherapy in the Treatment of Recurrent/Refractory Yolk Sac Tumor in Children
Acronym: SCRRYST
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shandong First Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HERO2020
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Germ Cell Tumor; Yolk Sac Tumor
Keywords: multiply relapsed or cisplatin refractory yolk sac tumor; sirolimus; germ cell tumor; mTOR
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Endodermal Sinus Tumor | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- sirolimus combined with chemotherapy treat recurrent/refractory yolk sac tumor in children (Experimental): This study employed an open single-group clinical laboratory design method (Simon Phase II study) to investigate the efficacy and safety of combining sirolimus with TIC chemotherapy (albumin-paclitaxel + isocyclophosphamide + carboplatin) in the treatment of children with recurrent/refractory vitellocystoma. AFP levels were assessed after each course of treatment, while imaging evaluations were conducted every two courses. The remission rate following chemotherapy in this single-group clinical trial was compared to that reported in the literature for treating recurrent/refractory yolk sac tumor, evaluating overall remission rate (ORR) and progresion-free survival rate (PFS) and overall survival (OS), as well as monitoring and recording chemotherapy-related side effects.
  Interventions: Drug: sirolimus combined with chemotherapy in the treatment of recurrent/refractory yolk sac tumor in children

INTERVENTIONS:
Drug: sirolimus combined with chemotherapy in the treatment of recurrent/refractory yolk sac tumor in children — The planned treatment protocol comprised four cycles of the S-TIC regimen, which included sirolimus administered orally at a dose of 1 mg/m² from day 1 to day 21-28, nab-paclitaxel at a dose of 200 mg/m² on day 1, ifosfamide at a dose of 1200 mg/m² from day 2 to day 5, and carboplatin at a dose of 400 mg/m² on day 2. Additionally, mesna and sulfamethoxazole were prescribed to prevent hemorrhagic cystitis and Pneumocystis Jirovecii Pneumonia (PJP), respectively. Each cycle spanned a duration of three to four weeks. AFP levels were evaluated at the end of each cycle, and radiological assessments were conducted every two cycles. Surgical intervention decisions were made based on the results of these assessments.

SUMMARY:
Remarkable progress has been made in treating germ-cell tumor (GCT) through the use of platinum-based regimens. However, part of yolk sac tumor (YST) with cisplatin resistance or recurrence is nevertheless prone to relapse after second-line treatment. This leaves a gap in effective treatment, which needs to be filled by novel therapeutic approaches. This paper is the first one to report the treatment combining sirolimus with nab-paclitaxel, ifosfamide, and carboplatin (S-TIC) for children with repeated relapsed or refractory yolk sac tumor (rrrYST).

DETAILED DESCRIPTION:
According to the latest relevant foreign case analysis reports and clinical trial results, the TIP regimen remains the recommended treatment for patients with recurrent and refractory malignant germ-cell tumors based on previous data. Carboplatin has been proven effective and less toxic in children with MGCTs, while cisplatin is more commonly used in early stages. In our research group's previously explored TIC scheme (albumin paclitaxel + ifosfamide + carboplatin), cisplatin is often substituted with carboplatin. Additionally, albumin paclitaxel replaces traditional paclitaxel due to its lower adverse reaction rate and higher tumor tissue uptake accumulation, forming the TIC regimen. Our preliminary clinical work has shown that the TIC regimen effectively improves remission rates of recurrent refractory germ cell tumors, particularly yolk sac tumors. For a small number of children who are not responsive to the TIC regimen, combining Sirolimus (an mTOR inhibitor) significantly enhances remission rates of recurrent refractory yolk sac tumors. This approach can potentially lead to cure or achieve surgery and radiotherapy within a curative timeframe. Therefore, this study aims to determine the efficacy of combining mTOR inhibitor Sirolimus with the TIC chemotherapy regimen (albumin-paclitaxel + isocyclophosphamide + carboplatin) in treating recurrent or refractory vitelline cyst tumors, providing a novel and effective therapeutic option for children with recurrent and refractory MGCTs.

ELIGIBILITY:
Inclusion Criteria：

* The pediatric patient is required to present histological confirmation of an extracranial yolk sac tumor.
* At the time of enrollment, the patient must be 18 years of age or younger, with no restrictions based on gender
* The patient must exhibit disease progression following a minimum of two platinum-based chemotherapy regimens or experience a relapse after the completion of treatment
* The patient must have measurable lesions, documented in accordance with the RECIST criteria, or possess an unassessable disease with alpha-fetoprotein (AFP) levels exceeding five times the upper limit of normal
* The Lansky performance status score must be 50 or higher, and the patient's life expectancy should be greater than 12 weeks
* The patient must have fully recovered from any prior adverse effects related to anti-cancer treatments

Exclusion Criteria：

* a history of previous tumors
* organ failure, specifically involving the heart, brain, liver, or kidneys.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
ORR: Objective Response Rate Allocation 'Non-Randomized' implies that this is a multi-arm study, but only one arm has been specified. Objective Response Rate | Each treatment cycle spans 3 to 4 weeks, 1-4 cycles, last at lest 3 to 16 weeks.
  Each treatment cycle spans 21 to 28 days (equivalent to every 3 to 4 weeks). Provided that the treatment criteria outlined in the study are satisfied, the second and subsequent cycles will commence on either the 22nd or 29th day. In the event of severe drug-related adverse reactions, treatment will be discontinued, and the patient will be classified as having PD. Tumor response assessment will entail the re-evaluation of AFP and LDH levels every cycle, alongside imaging examinations every two cycles. Should AFP levels demonstrate a continuous increase over two consecutive monitoring sessions following the initial treatment cycle, or if imaging results indicate tumor progression, a diagnosis of PD will be made, resulting in the termination of the clinical trial. For pediatric patients whose trials have been terminated, alternative anti-tumor therapies will be administered in accordance with their individual clinical conditions.

SECONDARY OUTCOMES:
Secondary endpoints included the progression-free survival (PFS) rate, overall survival (OS), and safety profile. | After each patient completed the clinical trial, they underwent imaging assessment examinations at 3/6/9/12/18/24/30/36/48/60 months after the end of the treatment.
  The study employed a Simon's two-stage optimal design with a one-sided alpha of 20% and 95% power to test the null hypothesis of ≤5% objective response rate (ORR) against the alternative hypothesis of ≥20% ORR. In the first stage, 10 patients were enrolled: if ≤1 patient achieved an objective response (CR/PR), the trial would be terminated for futility. Otherwise, enrollment would expand to a total of 32 patients. The regimen would be considered promising if ≥6 objective responses were observed in the final analysis. The median PFS and overall survival (OS) were estimated using the Kaplan-Meier method, implemented through the "survival" and "survminer" packages in R software (version 4.2.2). Correlations between OS and other endpoints were assessed at the patient level using Spearman's rank correlation coefficient (ρ).

CONTACTS AND LOCATIONS:
Overall Officials: Jingfu Wang, MD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No